CLINICAL TRIAL: NCT04775511
Title: Clinical and Ultrasonographic Comparison of the Effect of Hot and Cold Therapy on Spasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Banu Dilek, Assoc Prof, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DokuzUS
Record Dates: First submitted 2020-02-29; First posted 2021-03-01 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Spastic Hemiplegia
Keywords: spastisity; ultrasonography; hot pack; cold pack
MeSH Terms: conditions — Hemiplegia | interventions — Diathermy; Cryotherapy; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heat Therapy with heating pads (Experimental): 20 minutes of heating pads will be applied to the medial gastrocnemius muscle, followed by gastrocnemius muscle stretching for 20 minutes. While the patient is lying in a prone position the towel, which is located between the skin and heating pads, and heating pads will be placed on the gastrocnemius muscle.
  Interventions: Other: Heat Therapy with heating pads
- Cold Therapy with ice packs (Experimental): 20 minutes of ice packs will be applied to the medial gastrocnemius muscle, followed by gastrocnemius muscle stretching for 20 minutes. While the patient is lying in a prone position the towel, which is located between the skin and ice packs, and ice packs will be placed on the gastrocnemius muscle.
  Interventions: Other: Cold Therapy with ice packs
- Stretching Exercises (Other): 20 minutes of stretching exercises will be applied. In stretching exercises, stretching will be done for 30 seconds. The stretching exercises, which contain the maximal tension to the ankle, will be performed by the same physiotherapist while the patient is in the supine position, hip and knee extension.
  Interventions: Other: Stretching Exercises

INTERVENTIONS:
Other: Heat Therapy with heating pads — 20 minutes of heating pads will be applied to the medial gastrocnemius muscle, followed by gastrocnemius muscle stretching for 20 minutes. While the patient is lying in a prone position the towel, which is located between the skin and heating pads, and heating pads will be placed on the gastrocnemius muscle.
  Arms: Heat Therapy with heating pads
Other: Cold Therapy with ice packs — 20 minutes of ice packs will be applied to the medial gastrocnemius muscle, followed by gastrocnemius muscle stretching for 20 minutes. While the patient is lying in a prone position the towel, which is located between the skin and ice packs, and ice packs will be placed on the gastrocnemius muscle.
  Arms: Cold Therapy with ice packs
Other: Stretching Exercises — 20 minutes of stretching exercises will be applied. In stretching exercises, stretching will be done for 30 seconds. The stretching exercises, which contain the maximal tension to the ankle, will be performed by the same physiotherapist while the patient is in the supine position, hip and knee extension.
  Arms: Stretching Exercises

SUMMARY:
Spasticity is a positive sign of upper motor neuron syndrome. The frequency of spasticity development in patients with stroke is 38%. Spasticity is one of the important factors that negatively affect the rehabilitation potential and functional recovery of the patient. In the treatment of spasticity, oral antispasticide drugs, phenol, ethyl alcohol, botulinum toxin, and chemical nerve and motor point blocks, physical therapy, and rehabilitation, surgical methods are used. In the physical therapy rehabilitation program of spasticity, stretching and strengthening exercises, cold application, warm application, ultrasound therapy, electrical stimulation, biofeedback, extracorporeal shock therapy are used. Stretching exercises are the cornerstone of spasticity treatment. In many clinical and experimental studies, a decrease in spasticity has been noted after stretching exercises. It has been stated that the application of cold or hot applications before stretching may increase the effectiveness of spasticity treatment. The study comparing the effectiveness of hot and cold treatment applied before stretching exercises clinically and ultrasonographically has not been found in the literature. The purpose of this study is the evaluation of clinical and ultrasonographic comparison of the effect of hot and cold treatment on spasticity before stretching exercises in patients with stroke. This study is unique because it is the first study that evaluates the effect of hot and cold applications on spasticity before the stretching.

DETAILED DESCRIPTION:
The study is a randomized and controlled study. 30 patients will be included to study who apply to Dokuz Eylül University Faculty of Medicine, Department of Physical Medicine and Rehabilitation Clinic with the complaint of spasticity after stroke, aged between 18-75 years. These patients will be divided in three groups randomly (group1 n:10, group 2 n:10, group 3 n:10).

First group: 20 minutes of hot pack application to the medial gastrocnemius muscle. Then the patient will do stretching exercises to the gastrocnemius muscle, which will be done for 20 minutes. In hot pack for hot application; While the patient is lying in a prone position, a warm package, a towel between the skin and the skin will be applied on the gastrocnemius muscle and applied for 20 minutes.

Second group: 20 minutes to apply a cold pack to the medial gastrocnemius muscle, followed by stretching the patient for 20 minutes to the gastrocnemius muscle. The cold pack is available for cold application; While the patient is lying in a prone position, a cold pack will be placed on the gastrocnemius muscle, and a towel will be applied for 20 minutes.

Third group: 20 minutes of stretching and stretching exercises will be applied.

In stretching exercises, stretching will be done for 30 seconds. The stretching exercise will be performed by the same physiotherapist with maximal tension to the ankle in the supine position of the patient in the hip and knee extension.

These applications will continue as 5 sessions. Evaluations will be made before treatment, immediately after the first session and at the end of the 5th session. All patients will be evaluated for 3 times, before and after treatment and 5 session after the treatment with ultrasonographic measurements, ankle range of motion and spasticity degree.

Primary aim of this study is to evaluate the effect of hotpack and cold pack applicatios on Madial gastrokinemius ultrasonographic changes. For this purpose, medial muscle fascicule length, pennat angle and achilles tendon length with ultrasonographic measurement.

Secondary aim is evaluating the effect of hot and cold pack on spastisity and ankle range of motion. Spastisity will be measured by Aschwort scale and range of motion will be measured by goniomertry.

ELIGIBILITY:
Inclusion Criteria:

* Being first stroke attack
* Grade ≥1 Spasticity in the medial gastrocnemius muscle according to modified ashwort scale
* At least 6 weeks have passed since the stroke

Exclusion Criteria:

* Antispasticidal drug use
* Botulinum toxin injection into the gastrocnemius muscle
* Having another nervous system or orthopedic disease that can affect measurements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Medial gastrokinemius muscle via ultrasonographic measurement | All patients will be evaluated for 3 times; before treatment, first day of the treatment and fifth day of the treatment.
  Change of the medial gastrocinemius pennat angle, medial muscle fascicule length, achilles tendon length

SECONDARY OUTCOMES:
Change of the ankle range of motion | All patients will be evaluated for 3 times; before treatment, first day of the treatment and fifth day of the treatment.
  Ankle dorsiflexion will be measured by goniometry in knee extension and flexion.
Change of the degree of spastisity | All patients will be evaluated for 3 times; before treatment, first day of the treatment and fifth day of the treatment.
  Spastisity will be measured by Modified Aschwort Scale. (5 point numerical scale that graded spasticity from 0 to 4, with 0 being no resistance and 4 being a limb rigid in flexion or extension.)

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)